CLINICAL TRIAL: NCT00518076
Title: Staphylococcus Aureus Carriers Students Nursing Oxacillin Resistant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Other Study IDs: OF.262/2006-CEP
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2007-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Staphylococcal Infections
Keywords: Staphylococcus aureus carriers students nursing
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Staphylococcus aureus is an important pathogen bacteria actuating as an agent of a wide variety of infections, such as the superficials to the disseminates ones, its commonly find into hospitals ambient, assailing mainly immunosupress patients. Around 30% to 50% of people carries this agent in their nasal bone as part of their normal flora, occuring larger in hospitals workers. The S. aureus is also known for its high capacity of developing resistance to various antibiotic. Facing these considerations, the importance of nursing precaution and the infections control inside hospitals ambient, the purpose of this present study aimed to verify the rates of carriers of S. aureus in nursing students and the connection with the hospitals time involvement during graduation in the Faculty de Medicine de Botucatu - UNESP, embracing the 4 years of graduation college.

ELIGIBILITY:
Inclusion Criteria:

* Students nursing

Exclusion Criteria:

* Students nursing with infection

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Patrícia Pereira, Principal Investigator — São Paulo State University
Locations (1):
- São Paulo State University, Botucatu, São Paulo, Brazil